CLINICAL TRIAL: NCT01147289
Title: A Phase III, Randomized, Multicenter, Open Label Clinical Trial: Efficacy and Safety of the Injectable Association of Dexamethasone, Dipyrone, and Hydrocobalamin in Lumbar Sciatic Pain
Brief Title: Efficacy and Safety of Injectable Association of Dexamethasone, Dipyrone and Hydrocobalamin in Lumbar Sciatic Pain
Acronym: Dextra
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 102
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2012-05

CONDITIONS: Lumbar Sciatic Pain
Keywords: lumbar sciatic pain; moderate to severe lumbar sciatic pain within the last three days
MeSH Terms: interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexalgen (Experimental): Dexalgen® will be administered at a dose equivalent to dexamethasone 1.5 mg, dipyrone 500 mg, and hydroxocobalamin 5 mg (one ampoule for each type) a day at a single intramuscular dose for 3 days, at least
  Interventions: Drug: Dextralgen
- Meloxicam (Active Comparator): Meloxicam (Movatec®, Boehringer Ingelheim) will be administered as 15 mg (one ampoule) a day at a single intramuscular dose for at least 3 days.
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Dextralgen — Dexalgen® will be administered at a dose equivalent to dexamethasone 1.5 mg, dipyrone 500 mg, and hydroxocobalamin 5 mg (one ampoule for each type) a day at a single intramuscular dose. Both drugs will be administered for 3 days, at least.
  Arms: dexalgen
Drug: Meloxicam — Meloxicam (Movatec®, Boehringer Ingelheim) will be administered as 15 mg (one ampoule) a day at a single intramuscular dose. Both drugs will be administered for 3 days, at least.
  Arms: Meloxicam

SUMMARY:
A phase III, randomized, multicenter, open label clinical trial to evaluate efficacy and safety of the injectable association of dexamethasone, dipyrone, and hydroxocobalamin in lumbar sciatic pain. The study will enroll 140 patients in each arm (280 total).

ELIGIBILITY:
Inclusion Criteria:

* Sign the study informed consent form;
* To be diagnosed with moderate to severe lumbar sciatic pain (defined as limiting the work activities or the ordinary tasks performance or at the investigator's discretion) within the last 3 days;
* Aged 18 to 75 years old;
* To be able to meet the study procedures

Exclusion Criteria:

o-Diagnosed with chronic rheumatologic diseases, except recurrent lumbar sciatic pain;

* Patients with one of the following conditions, as per the investigator's criteria:
* Severe renal failure under hemodialysis, severe liver failure, uncontrolled severe heart failure;
* Severe injuries on gastrointestinal tract;
* Other severe comorbidities;
* Patients taking acetylsalicylic acid or any anti-clotting;
* Female patients who are pregnant, lactating, willing to get pregnant or not willing to use an appropriate contraceptive method during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
efficacy | 6 months
  The efficacy analysis will be at the per protocol population, with the VAS measure after three treatment dosages. The VAS scale consists on a straight line of 100 mm in which the patient marks, at any point through the straight line, the point he/she considers to describe the pain level he/she feels. After the patient marks the straight line, classifying his/her pain, it is measured with a millimeter-graded standard rule, the distance between the mark and the extremity "No pain" at the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gorios, Phd./MD, Principal Investigator — Sociedade Beneficente São Camilo; Paulo Guilherme Oliveira e Silva, Phd/MD, Principal Investigator — Hospital Santa Marcelina; Luciana Teixeira Pinto, Phd/MD, Principal Investigator — Instituto de Pesquisa Clínica e Medicina Avançada (IMA); Sergio Raj Eis, Phd/MD, Principal Investigator — CEDOES; Jose Alexandre Mendonça, Phd/MD, Principal Investigator — Instituto de Pesquisa Clínica de Campinas (IPECC); Sonia Maria Silva, Phd/MD, Principal Investigator — Faculdade de Medicina ABC
Locations (6):
- Brazil (6):
  - CEDOES, Vitória, Espírito Santo
  - Sociedade Beneficente São Camilo, Campinas, São Paulo
  - Instituto De Pesquisa Clínica De Campinas IPECC, Campinas, São Paulo
  - Instituto de Pesquisa Clínica e Medicina Avançada Ltda IMA, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Faculdade de Medicina ABC, São Paulo, São Paulo